CLINICAL TRIAL: NCT01295255
Title: Interaction Effect of Asthma and Aeroallergen Category on the Psychological Status in Allergic Rhinitis Patients
Status: Completed | Type: Observational
Sponsor: Beijing Tongren Hospital (Other)
Responsible Party: Demin Han, Beijing Tongren Hospital
Other Study IDs: 1130
Record Dates: First submitted 2011-02-11; First posted 2011-02-14 (Estimated); Last update posted 2011-02-14 (Estimated); Status verified 2011-01

CONDITIONS: Hypersensitivity; Psychologic Factors in Physical Conditions Classified Elsewhere; Respiratory Tract Diseases; Allergic Rhinitis
Keywords: Allergic rhinitis; Psychological status; Asthma; Aeroallergen
MeSH Terms: conditions — Hypersensitivity; Respiratory Tract Diseases; Rhinitis, Allergic; Asthma

STUDY DESIGN:
Observational Model: Cohort

SUMMARY:
Allergic rhinitis (AR) and asthma are considered as "one airway, one disease". Although there is increasing evidence for an association between allergy and depression, it remains unknown if the relationship between AR and asthma has extra influence on the psychological status of the patients. The aim of our study was to investigate the influence pattern of asthma on the psychological status in AR patients. The Symptom Checklist-90 (SCL-90) was employed to analyze the psychological status of 524 individuals with AR. Independent sample T-tests, one-way ANOVA and multivariate ANOVA were used for data analyses.

ELIGIBILITY:
Inclusion Criteria:

* Patients suffered from rhinitis symptoms such as nasal itching, sneezing, nasal obstruction and running nose, all patients had not undergone any medicine therapy in the past one week; nasal endoscopy showed a pale and edematous nasal mucosa, nasal discharge and swollen inferior turbinates. Every nasal symptom was scored on Visual analog scale (VAS, 0-3 score) respectively. A score of 0 indicated no nasal symptom, 1 indicated slight nasal symptoms, 2 indicated obvious nasal symptom, but which could still be endured, and 3 indicated obvious nasal symptoms that could not be endured;
* Age between 16 to 60 years;
* A positive skin prick test (SPT)to at least one allergen, the level of response equal to or exceeding ++. The following inhalant allergens were tested: Der p; Der f; Animal hair; Trees; Grasses; Cereals; Mugwort; Dandelion; Giant ragweed; Chenopodium album; Humulus; Locust; Blatella germanica; Pine; Plantain; Curvularia lunata; Candida albicans; Penicillium notatum; Alternaria tenuis and Aspergillus fumigatu. The reactions were evaluated based on the mean wheal diameter at 15 minutes after application of the extracts. The mean diameters of each allergen wheals were calculated from the sum of the largest measurement across the wheal and the largest wheal measurement perpendicular to this divided by two. In addition, we calculated the skin index (SI) as the ratio of allergen weal diameter divided by the histamine weal size. The SPT result for each allergen was defined in terms of the SI value as follows: +: SI≤0.5; ++: 0.5<SI≤1.0; +++: 1.0<SI≤2.0; ++++: SI>2.0.

Exclusion Criteria:

* AR combined with hypertension, diabetes or other chronic diseases;
* AR combined with tumor in the nasal cavity;
* AR combined with eczema;
* Acute infection in the past one week;
* Failure to complete the questionnaires;
* AR patients undergoing negative life events.

Ages: 16 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: 524 affected individuals (311 males and 213 females) with AR were prospectively recruited from the rhinology clinic of the Otolaryngology, Head and Neck Surgery Department of Beijing Tongren Hospital from February 2009 to November 2009.
Sampling Method: Probability Sample
Enrollment: 524 (Actual)
Dates: Start 2009-02; Primary Completion 2009-10 (Actual); Study Completion 2009-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: DeMin Han, Phd, Principal Investigator — Beijing Tongren Hospital